CLINICAL TRIAL: NCT02993627
Title: Effects of Spirulina Supplementation on Anthropometric Measurements, Lipid Profile, Appetite, Liver Enzymes, Inflammatory and Glycemic Markers on Overweight or Obese Adults
Brief Title: Effects of Spirulina Supplementation on Overweight or Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Atoosa Saidpour, Assistant Professor of Nutrition Science, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.nnftri.Rec.1395.63
Record Dates: First submitted 2016-11-27; First posted 2016-12-15 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: obesity; BMI; body weight
MeSH Terms: conditions — Obesity; Body Weight | interventions — Diet Therapy; Diet, Reducing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spirulina (Experimental): daily intake of spirulina tablets weight reduction diet therapy
  Interventions: Dietary Supplement: Spirulina; Other: diet therapy
- placebo (Placebo Comparator): daily intake of placebo tablets weight reduction diet therapy
  Interventions: Other: diet therapy

INTERVENTIONS:
Dietary Supplement: Spirulina — 2 g(4* 500 mg tablets) daily intake of Spirulina Platensis
  Other Names: Spiruvit
  Arms: Spirulina
Other: diet therapy — low calorie diet (-500 or -300 kcal) composed of 55% carbohydrate, 15% protein and 30% fat
  Other Names: weight reduction diet

SUMMARY:
In this double-blind Randomized Controlled Clinical Trial investigators are going to study the effects of Spirulina supplementation on anthropometric measurements, lipid profile, appetite, liver enzymes, inflammatory and glycemic markers in a sample of overweight or obese adults.

DETAILED DESCRIPTION:
A sample of 40 obese and overweight subjects will be recruited from Nutrition And Diet Therapy Clinic Of Shahid Beheshti Medical University.

This study is a double-blind Randomized Controlled Clinical Trial, that subjects will be randomly allocated to spirulina or placebo group according to the Random permuted blocks within strata method based on BMI. Subjects will consume 2 g spirulina daily (4 tablets of 500mg), whereas the control group are going to receive identical placebo tablets. Subjects are asked to maintain their usual physical activity level during the intervention period and also avoid taking any other supplements or medications without consulting the investigators. Intervention period is designed to be 12 weeks that has been determined sufficient to record changes of study parameters. At the beginning of the study and after 12 weeks of intervention, morning blood samples will be collected after 12 h of fasting. Anthropometric parameters will be also measured at the beginning, week 6 and after 12 weeks of intervention. Subjects will be followed through social network to ensure their compliance with the study. Furthermore, subjects in both spirulina and placebo groups received low calorie diet (-500 or -300 kcal) composed of 55% carbohydrate, 15% protein and 30% fat during the study period.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25 kg/m2
* No history of medications for obesity, diabetes, dyslipidemia, inflammatory disease within 3 months before the study
* No history of vitamin or antioxidant supplementation within 3 months before the study
* Giving written informed consent for participation

Exclusion Criteria:

* Having chronic kidney or hepatic disease except NAFLD
* Havig hypo or hyperthyroidism
* Having autoimmune and infectious disease
* weight reduction diet therapy within 6 month from the intervention
* Having more than 3kg weight change in recent 2 months
* Having recent surgery
* Taking anticoagulant drugs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
body weight | week 12
  body weight with minimum of clothes and without shoes through a calibrated scale and with the precision of 100gr
BMI | week 12
  calculation
waist circumference | week 12
  measuring with an inflexible tapeline with the precision of 0.1cm
hip circumference | week 12
  measuring with an inflexible tapeline with the precision of 0.1cm
waist/hip ratio | week 12
  calculation
body fat mass | week 12
  bioempedance
body fat free mass | week 12
  bioempedance
apetite | week 12
  questionaire

SECONDARY OUTCOMES:
serum triaylglycerol | week 12
  enzymatic method
serum total cholesterol | week 12
  enzymatic method
e serum HDL-C | week 12
  enzymatic method
serum LDL-C | week 12
  calculation
serum LDL-C/HDL-C | week 12
  calculation
serum fasting glucose | week 12
  enzymatic method
serum insulin | week 12
  enzymatic method
HOMA-IR | week 12
  calculation
serum hs-CRP | week 12
  eliza
serum adiponectin | week 12
  eliza
serum SGOT | week12
  enzymatic method
serum SGPT | week 12
  enzymatic method

CONTACTS AND LOCATIONS:
Overall Officials: Atoosa Saidpour, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Clinical Nutrition and Diet Therapy Clinic of Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torres-Duran PV, Ferreira-Hermosillo A, Juarez-Oropeza MA. Antihyperlipemic and antihypertensive effects of Spirulina maxima in an open sample of Mexican population: a preliminary report. Lipids Health Dis. 2007 Nov 26;6:33. doi: 10.1186/1476-511X-6-33. PMID 18039384
- [Result] Park HJ, Lee YJ, Ryu HK, Kim MH, Chung HW, Kim WY. A randomized double-blind, placebo-controlled study to establish the effects of spirulina in elderly Koreans. Ann Nutr Metab. 2008;52(4):322-8. doi: 10.1159/000151486. Epub 2008 Aug 19. PMID 18714150
- [Result] Parikh P, Mani U, Iyer U. Role of Spirulina in the Control of Glycemia and Lipidemia in Type 2 Diabetes Mellitus. J Med Food. 2001 Winter;4(4):193-199. doi: 10.1089/10966200152744463. PMID 12639401
- [Result] Miczke A, Szulinska M, Hansdorfer-Korzon R, Kregielska-Narozna M, Suliburska J, Walkowiak J, Bogdanski P. Effects of spirulina consumption on body weight, blood pressure, and endothelial function in overweight hypertensive Caucasians: a double-blind, placebo-controlled, randomized trial. Eur Rev Med Pharmacol Sci. 2016;20(1):150-6. PMID 26813468
- [Result] Mazokopakis EE, Papadomanolaki MG, Fousteris AA, Kotsiris DA, Lampadakis IM, Ganotakis ES. The hepatoprotective and hypolipidemic effects of Spirulina (Arthrospira platensis) supplementation in a Cretan population with non-alcoholic fatty liver disease: a prospective pilot study. Ann Gastroenterol. 2014;27(4):387-394. PMID 25331487
- [Result] Lee EH, Park JE, Choi YJ, Huh KB, Kim WY. A randomized study to establish the effects of spirulina in type 2 diabetes mellitus patients. Nutr Res Pract. 2008 Winter;2(4):295-300. doi: 10.4162/nrp.2008.2.4.295. Epub 2008 Dec 31. PMID 20016733
- Available data/document: Clinical Study Report: 18039384 — http://lipidworld.biomedcentral.com/articles/10.1186/1476-511X-6-33/